CLINICAL TRIAL: NCT04598698
Title: Endometriosis Diagnosis Using MicroRNA: Prospective Study in Women to Allow Early Disease Recognition
Brief Title: The EMPOWER Study: Endometriosis Diagnosis Using MicroRNA
Acronym: EMPOWER
Status: Active, not recruiting | Type: Observational
Sponsor: Dot Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Dot Laboratories DL-001
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Endometriosis is a complex, heterogeneous disease that may present inconsistently across women. Using disease-specific biomarkers and advanced biostatistics, DotLab is developing a biomarker test to confirm the presence of endometriosis.This is a multi-center, prospective, observational, minimal risk study in women undergoing laparoscopy, laparotomy or other pelvic surgical procedure for endometriosis, infertility or another benign gynecological indication. Participants will undergo 2 study visits for collection of blood and saliva and completion of study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to provide written informed consent.
2. Participant is willing and able to provide up to 50 mL of blood via venipuncture and comply with all other study and sample collection procedures.
3. Participant is a female aged 18 through 49 years (inclusive).
4. Participant is scheduled to undergo:

   1. Laparotomy or laparoscopy for signs and symptoms of suspected endometriosis. This shall constitute approximately 95% of the participants enrolled.
   2. Laparotomy, laparoscopy, or other procedures including, but not limited to, tubal ligation, lysis of adhesions, hysterectomy for benign condition, myomectomy, salpingo-oophorectomy, cystectomy, or diagnostic laparoscopy for indications including, but not limited to, infertility or benign gynecological indications (e.g., benign pelvic masses, infertility, abnormal uterine bleeding). This shall constitute approximately 5% of the participants enrolled.

Exclusion Criteria:

1. Participant has a history of surgically determined diagnosis of endometriosis (either via visual inspection or histopathology).
2. Participant is a female in a pre-menarchal or post-menopausal state (last menstrual period at least 1 year before Screening and no other biological or physiological cause can be identified) or has been rendered surgically menopausal (bilateral oophorectomy) for at least 6 months at Screening.
3. Participant is pregnant.
4. Participant has an active malignancy.
5. Participant is known to have tested positive for human immunodeficiency virus or hepatitis A, B, or C.
6. Participant has an active pelvic infection or other infections contraindicated for surgery.
7. Participant has participated (±3 months of study enrollment) in a clinical trial where an investigational drug was or is planned to be administered.
8. Participant has any general health or behavioral condition that, in the opinion of the investigator, should exclude the participant from participation.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women of reproductive age who have been referred to surgery for suspected endometriosis and other benign gynecological indications.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical validity | From date of first sample collection to surgery, up to 3 weeks
  Performance of a microRNA (miRNA)-based assay compared to visual inspection during surgery for the diagnosis of active endometriosis

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Stanford University Hospital, Palo Alto, California
  - Center for Special Minimally Invasive & Robotic Surgery, Woodside, California
  - Yale University, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - RAD Fertility, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Academia of Women's Health and Endoscopic Surgery, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - The Advanced Gynecologic Surgery Institute, Park Ridge, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Rutgers Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - NewYork-Presbyterian / Columbia University Medical Center, New York, New York
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Health, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Austin, Austin, Texas
  - Seattle Reproductive Medicine, Seattle, Washington